CLINICAL TRIAL: NCT03621501
Title: Percutaneous Complete Revascularization Strategies Using Sirolimus Eluting Biodegradable Polymer Coated Stents in Patients Presenting With Acute Coronary Syndrome and Multivessel Disease
Brief Title: Direct Complete Versus Staged Complete Revascularization in Patients Presenting With Acute Coronary Syndromes and Multivessel Disease
Acronym: BioVasc
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Principal Investigator, Roberto Diletti, Dr., Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BioVasc protocol definitive
Record Dates: First submitted 2018-02-08; First posted 2018-08-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Percutaneous coronary intervention; Multivessel disease
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicenter, randomized, two-arm, international, open-label, non-inferiority study. Due to the design characteristics of the study, the study investigators and operators cannot be blinded.
Who Masked: Outcomes Assessor
Masking Description: The clinical event adjudication committee, consisting of cardiologists who are not participating in the study, will be blinded for the treatment arm of the patients to avoid a potential bias in the adjudication process of events
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staged complete revascularization (Placebo Comparator): • Culprit only + staged (within six weeks after index procedure) complete revascularization in all vessels ≥ 2.5mm with ≥ 70% stenosis by visual estimation or positive coronary physiology test per operator's discretion (Control arm)
  Interventions: Device: Percutaneous coronary intervention
- Immediate complete revascularization (Active Comparator): • Immediate complete revascularization in all vessels ≥ 2.5mm with ≥ 70% stenosis by visual estimation or positive coronary physiology test per operator's discretion (Experimental arm)
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — At the index procedure, the culprit lesion (cause of complaints/acute coronary syndrome) will be treated according to standard of care with a Biotronik Orsiro DES (Sirolimus-Eluting stent). If there are additional significant lesions besides the culprit lesion, patients will be randomized to direct complete revascularization or staged complete revascularization. In the direct complete revascularization group all lesions will be treated during the index procedure. In the staged complete revascularization group, only the culprit lesion will be treated during the index procedure. The remaining significant lesions will be treated later but within six weeks after the index procedure. In both arms the additional lesions will also be treated with Biotronik Orsiro DES (Sirolimus-Eluting stent).
  Other Names: PCI

SUMMARY:
To test whether immediate complete revascularization is non-inferior to staged (but within six weeks after index procedure) complete revascularization in Patients presenting with ACS, including Non-ST-elevation ACS (NSTEACS) and ST-elevation myocardial infarction (STEMI), with multivessel disease accepted for PCI

DETAILED DESCRIPTION:
Invasive coronary angiography followed by percutaneous coronary intervention is the treatment of choice in patient presenting with STEMI-ACS1 and NSTE-ACS2. Up to 60 percent of these patients have multivessel disease on angiography3-5. Patients with multivessel disease have a worse prognosis compared with patients having culprit vessel disease only5. It has been debated whether a complete or culprit artery only revascularization strategy is better.

Retrospective data in STEMI patients suggested a lower mortality in patients that were treated with culprit artery only compared with multivessel PCI during index procedure6. Since then, four randomized controlled trials have addressed this question in STEMI population; The Randomized Trial of Preventive Angioplasty in Acute Myocardial Infarction (PRAMI) trial (n = 465, 23 months follow-up)7, the Randomized trial of complete versus lesion-only revascularization in patients undergoing primary percutaneous coronary intervention for STEMI and multivessel disease (CvLPRIT) (n = 296, 12months follow-up)8, the Complete revascularisation versus treatment of the culprit lesion only in patients with ST-segment elevation myocardial infarction and multivessel disease (DANAMI-3-PRIMULTI) trial (n = 627, 27months follow-up)9, and the Fractional Flow Reserve-Guided Multivessel Angioplasty in Myocardial Infarction (Compare-Acute) trial (n = 885, 12 months follow-up)10. PCI of the non-infarct related artery was performed at the index procedure (PRAMI and Compare-Acute), staged before discharge (DANAMI-3-PRIMULTI) or at any time during hospitalization (CvLPRIT). Indication for PCI was significant stenosis as assessed by angiography (PRAMI and CvLPRIT) or FFR (DANAMI-3-PRIMULTI and COMPARE-ACUTE). There was a significant reduction in primary outcome in all four trials in favor of complete revascularization. However, there was no significant reduction in total mortality or myocardial infarction. Based on the results for these four trials, the 2017 ESC STEMI-ACS guidelines gave a class II, level of evidence (LOE) A, indication for routine complete revascularization in STEMI patients with multivessel disease, including those presenting with cardiogenic shock1. However, an important shortcoming of the abovementioned studies is the absence of a staged complete revascularization arm. As there is no data that compare immediate and staged complete revascularization, the guidelines don't advise on when to perform non-infarct related artery revascularization.

Data regarding optimal treatment in NSTEMI-ACS are more scarce. In an observational study by Shishesbor and coworkers, they showed that nonculprit multivessel stenting reduced future revascularization rate but this was not associated with lower rate of death or myocardial infarction11. Recently, a substudy from the Bleeding complications in a Multicenter registry of patients discharged with diagnosis of acute coronary syndrome (BleeMACS) registry (N=4520 patients, 1459 NSTEMI) was published12. They showed that in NSTEMI patients, complete revascularization was associated with a significant lower rate of death (4.5% vs. 8.5%; p=0.002), re-AMI (3.7% vs. 6.6%; p=0.016) and MACE (8.1% vs. 13.9%; p=0.001) at one year follow up. The 2015 ESC NSTEMI-ACS guidelines not specifically advise a culprit only or multivessel PCI strategy. Moreover, they advise to base revascularization strategy on patients clinical status and co-morbidities, as well as disease severity, Class II, LEO B. Interestingly, in contrast with the STEMI population, in NSTEMI population there is a small RCT investigating staged versus direct complete revascularization , the Single-Staged Compared With Multi-Staged PCI in Multivessel NSTEMI Patients: The SMILE Trial (N=584 patients)13. There was a significant reduction in primary endpoint 1S-PCI: n = 36 [13.63%] vs. MS-PCI: n = 61 [23.19%]; hazard ratio [HR]: 0.549 [95% confidence interval (CI): 0.363 to 0.828]; p = 0.004) at one year follow up. This was mainly driven by a reduction in target vessel revascularization. There was no significant difference in cardiac death or myocardial infarction between the both groups. This finding deserves further investigation, because the TVR rate (15.4% at 1 year) in the multistage group was unprecedentedly high in the era of current-generation drug-eluting stents.

There is no publication specifically addressing the patients with unstable angina regarding the subject of complete or incomplete revascularization or timing of revascularization.

Considering such data, complete revascularization in ACS patients seems advisable, but timing of revascularization is unknown.

Given this background no investigation so far provided a comprehensive evaluation of the complete revascularization strategies for patients with any type of acute coronary syndrome and multivessel disease. Therefore, the investigators aim to investigate in a randomized controlled trial the commonly used complete revascularization strategies for patients presenting with ACS: 1) Immediate complete revascularization 2) Culprit only plus staged complete revascularization within six weeks after index procedure, in terms of the primary endpoint, the composite of death from any cause, nonfatal type 1 myocardial infarction, revascularization, and cerebrovascular events at 1-year post intervention.

Patients will be treated with one commercially available second-generation drug-eluting stent stent to ensure homogeneity of treatment among patients, abolishing the occurrence of bias due to different stent usage. The stents used will be the Biotronik Orsiro DES (Sirolimus-Eluting stent). The Orsiro DES is a second generation DES with a bioabsorbable polymer coating releasing sirolimus and was CE marketed in 2011. The bioabsorbable nature of the polymer could be associated with a reduction of the inflammatory response, reducing neo-intima growth compared to a durable polymer14, 15. The active drug sirolimus is a lipophilic molecule that inhibits mammalian target of rapamycine (mTOR) on smooth muscle cells, also preventing neo-intima hyperplasia16. The Orsiro stent has ultrathin cobalt chromium struts of 60-80micron (depending on stent size) enhancing deliverability and crossability without loss of radial strength or fatigue resistance. The Orsiro stent has been extensively studied in different study populations with more than 32.500 patients studied globally.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria STEMI-ACS ST-segment elevation myocardial infarction (STEMI) Both criteria must be present for eligibility

* Chest pain for more than 20 minutes with an electrocardiographic ST-segment elevation of 1 mm or greater in two or more contiguous leads, or with a new left bundle-branch block
* Admission either within 12 hours of symptom onset or between 12 and 24 hours after onset with evidence of continuing ischemia.

Inclusion criteria for NSTE-ACS Non-ST-segment elevation myocardial infarction (NSTEMI) At least two of the following must be present for eligibility

* History consistent with new, or worsening ischemia, occurring at rest or with minimal activity
* Coronary angiography with indication to PCI
* Troponin T or I or creatine kinase MB above the upper limit of normal
* Electrocardiographic changes compatible with ischemia but not diagnostic for ST-segment elevation myocardial infarction (i.e. ST depression of 1 mm or greater in two contiguous leads, T-wave inversion more than 3 mm, or any dynamic ST shifts) 0 Unstable Angina (UA)

At least two of the following must be present in the absence of cardiomyocyte necrosis (i.e. Troponin T or I and creatine kinase MB must be within normal limits):

* History consistent with new, or worsening ischemia, occurring at rest or with minimal activity
* Coronary angiography with indication to PCI
* Electrocardiographic changes compatible with ischemia but not diagnostic for ST-segment elevation myocardial infarction (i.e. ST depression of 1 mm or greater in two contiguous leads, T-wave inversion more than 3 mm, or any dynamic ST shifts)

General inclusion criteria:

* Age ≥ 18 years ≤ 85 years
* The patient is an acceptable candidate for treatment with a drug eluting stent in accordance with the applicable guidelines on percutaneous coronary interventions, manufacturer's Instructions for Use and the Declaration of Helsinki
* Patient indication, lesion length and vessel diameter of the target lesion(s) are according to the 'Instructions for Use' that comes with every Biotronik Orsiro (Sirolimus-Eluting stent) system.
* The patient is willing and able to cooperate with study procedures and the required follow up visits
* The subject or legal representative has been informed of the nature of the study and agrees to its provisions and has provided an EC approved written informed consent, including data privacy authorization

Exclusion Criteria:

* Age <18 years and > 85 years
* Single coronary vessel disease or multivessel disease without clear culprit
* Patients in cardiogenic shock
* Patients who cannot give informed consent or have a life expectancy of less than 1year
* Absolute contraindications or allergy that cannot be pre-medicated, to iodinated contrast or to any of the study medications, including both aspirin and P2Y12 inhibitors.
* Enrollment in another study with another investigational device or drug trial that has not reached the primary endpoint . The patient may only be enrolled once in the BioVAsc study
* PCI in the previous 30 days.
* Presence of a chronic total occlusion
* Previous CABG
* Women of childbearing potential who do not have a negative pregnancy test within 7 days before the procedure and women who are breastfeeding.
* Planned surgery within 6 months after PCI, unless dual antiplatelet therapy is maintained throughout the peri-surgical period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1525 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
MACCE | 1 year
  a composite clinical outcome of all-cause mortality, myocardial infarction, any unplanned ischemia driven revascularization, and cerebrovascular events

SECONDARY OUTCOMES:
MACCE | 30 days
  Composite clinical outcome of all-cause mortality, myocardial infarction, any unplanned ischemia driven revascularization, and cerebrovascular events
MACCE | 2 years
  Composite clinical outcome of all-cause mortality, myocardial infarction, any unplanned ischemia driven revascularization, and cerebrovascular events
MACCE | 5 years
  Composite clinical outcome of all-cause mortality, myocardial infarction, any unplanned ischemia driven revascularization, and cerebrovascular events
All cause mortality | 30 days
  All cause mortality
All cause mortality | 1 year
  All cause mortality
All cause mortality | 2 years
  All cause mortality
All cause mortality | 5 years
  All cause mortality
Myocardial infarction | 30 days
  Myocardial Infarction
Myocardial infarction | 1 year
  Myocardial Infarction
Myocardial infarction | 2 years
  Myocardial Infarction
Myocardial infarction | 5 years
  Myocardial Infarction
Coronary revascularization | 30 days
  Any unplanned ischemia driven coronary revascularization procedure
Coronary revascularization | 1 year
  Any unplanned ischemia driven coronary revascularization procedure
Coronary revascularization | 2 years
  Any unplanned ischemia driven coronary revascularization procedure
Coronary revascularization | 5 years
  Any unplanned ischemia driven coronary revascularization procedure
Major bleeding | 30 days
  Major bleeding (not related to coronary-artery bypass grafting, BARC 3-5)
Major bleeding | 1 year
  Major bleeding (not related to coronary-artery bypass grafting, BARC 3-5)
Need for renal replacement therapy | 30 days
  Need for renal replacement therapy
Quality of Life Seattle Angina Questionnaire | 30 days
  Seattle Angina Questionnaire. Scale 1-5. Higher values represent better outcome
Quality of life Seattle Angina Questionnaire | 1 year
  Seattle Angina Questionnaire. Scale 1-5. Higher values represent better outcome
Quality of Life EQ5D | 30 days
  EQ5D EQ5D EQ5D. Scale 1-5. Higher values represent worse outcome
Quality of life EQ5D | 1 year
  EQ5D. Scale 1-5. Higher values represent worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Diletti, Dr., Principal Investigator — Erasmus Medical Center; Nicolas Van Mieghem, Prof., Study Chair — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Result] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Result] D'Ascenzo F, Presutti DG, Picardi E, Moretti C, Omede P, Sciuto F, Novara M, Yan AT, Goodman S, Mahajan N, Kosuge M, Palazzuoli A, Jong GP, Isma'eel H, Budoff MJ, Rubinshtein R, Gewirtz H, Reed MJ, Theroux P, Biondi-Zoccai G, Modena MG, Sheiban I, Gaita F. Prevalence and non-invasive predictors of left main or three-vessel coronary disease: evidence from a collaborative international meta-analysis including 22 740 patients. Heart. 2012 Jun;98(12):914-9. doi: 10.1136/heartjnl-2011-301596. PMID 22626899
- [Result] Fox KA, Poole-Wilson PA, Henderson RA, Clayton TC, Chamberlain DA, Shaw TR, Wheatley DJ, Pocock SJ; Randomized Intervention Trial of unstable Angina Investigators. Interventional versus conservative treatment for patients with unstable angina or non-ST-elevation myocardial infarction: the British Heart Foundation RITA 3 randomised trial. Randomized Intervention Trial of unstable Angina. Lancet. 2002 Sep 7;360(9335):743-51. doi: 10.1016/s0140-6736(02)09894-x. PMID 12241831
- [Result] Park DW, Clare RM, Schulte PJ, Pieper KS, Shaw LK, Califf RM, Ohman EM, Van de Werf F, Hirji S, Harrington RA, Armstrong PW, Granger CB, Jeong MH, Patel MR. Extent, location, and clinical significance of non-infarct-related coronary artery disease among patients with ST-elevation myocardial infarction. JAMA. 2014 Nov 19;312(19):2019-27. doi: 10.1001/jama.2014.15095. PMID 25399277
- [Result] Hannan EL, Samadashvili Z, Walford G, Holmes DR Jr, Jacobs AK, Stamato NJ, Venditti FJ, Sharma S, King SB 3rd. Culprit vessel percutaneous coronary intervention versus multivessel and staged percutaneous coronary intervention for ST-segment elevation myocardial infarction patients with multivessel disease. JACC Cardiovasc Interv. 2010 Jan;3(1):22-31. doi: 10.1016/j.jcin.2009.10.017. PMID 20129564
- [Result] Wald DS, Morris JK, Wald NJ, Chase AJ, Edwards RJ, Hughes LO, Berry C, Oldroyd KG; PRAMI Investigators. Randomized trial of preventive angioplasty in myocardial infarction. N Engl J Med. 2013 Sep 19;369(12):1115-23. doi: 10.1056/NEJMoa1305520. Epub 2013 Sep 1. PMID 23991625
- [Result] Gershlick AH, Khan JN, Kelly DJ, Greenwood JP, Sasikaran T, Curzen N, Blackman DJ, Dalby M, Fairbrother KL, Banya W, Wang D, Flather M, Hetherington SL, Kelion AD, Talwar S, Gunning M, Hall R, Swanton H, McCann GP. Randomized trial of complete versus lesion-only revascularization in patients undergoing primary percutaneous coronary intervention for STEMI and multivessel disease: the CvLPRIT trial. J Am Coll Cardiol. 2015 Mar 17;65(10):963-72. doi: 10.1016/j.jacc.2014.12.038. PMID 25766941
- [Result] Engstrom T, Kelbaek H, Helqvist S, Hofsten DE, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Clemmensen P, De Backer O, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Kober L; DANAMI-3-PRIMULTI Investigators. Complete revascularisation versus treatment of the culprit lesion only in patients with ST-segment elevation myocardial infarction and multivessel disease (DANAMI-3-PRIMULTI): an open-label, randomised controlled trial. Lancet. 2015 Aug 15;386(9994):665-71. doi: 10.1016/s0140-6736(15)60648-1. PMID 26347918
- [Result] Smits PC, Abdel-Wahab M, Neumann FJ, Boxma-de Klerk BM, Lunde K, Schotborgh CE, Piroth Z, Horak D, Wlodarczak A, Ong PJ, Hambrecht R, Angeras O, Richardt G, Omerovic E; Compare-Acute Investigators. Fractional Flow Reserve-Guided Multivessel Angioplasty in Myocardial Infarction. N Engl J Med. 2017 Mar 30;376(13):1234-1244. doi: 10.1056/NEJMoa1701067. Epub 2017 Mar 18. PMID 28317428
- [Result] Shishehbor MH, Lauer MS, Singh IM, Chew DP, Karha J, Brener SJ, Moliterno DJ, Ellis SG, Topol EJ, Bhatt DL. In unstable angina or non-ST-segment acute coronary syndrome, should patients with multivessel coronary artery disease undergo multivessel or culprit-only stenting? J Am Coll Cardiol. 2007 Feb 27;49(8):849-54. doi: 10.1016/j.jacc.2006.10.054. Epub 2007 Feb 8. PMID 17320742
- [Result] Quadri G, D'Ascenzo F, Moretti C, D'Amico M, Raposeiras-Roubin S, Abu-Assi E, Henriques JPS, Saucedo J, Gonzalez-Juanatey JR, Wilton SB, Kikkert WJ, Nunez-Gil I, Ariza-Sole A, Song X, Alexopoulos D, Liebetrau C, Kawaji T, Huczek Z, Nie SP, Fujii T, Correia L, Kawashiri MA, Garcia-Acuna JM, Southern D, Alfonso E, Terol B, Garay A, Zhang D, Chen Y, Xanthopoulou I, Osman N, Mollmann H, Shiomi H, Omede P, Montefusco A, Giordana F, Scarano S, Kowara M, Filipiak K, Wang X, Yan Y, Fan JY, Ikari Y, Nakahashi T, Sakata K, Yamagishi M, Kalpak O, Kedev S, Varbella F, Gaita F. Complete or incomplete coronary revascularisation in patients with myocardial infarction and multivessel disease: a propensity score analysis from the "real-life" BleeMACS (Bleeding complications in a Multicenter registry of patients discharged with diagnosis of Acute Coronary Syndrome) registry. EuroIntervention. 2017 Jul 20;13(4):407-414. doi: 10.4244/EIJ-D-16-00350. PMID 28169217
- [Result] Sardella G, Lucisano L, Garbo R, Pennacchi M, Cavallo E, Stio RE, Calcagno S, Ugo F, Boccuzzi G, Fedele F, Mancone M. Single-Staged Compared With Multi-Staged PCI in Multivessel NSTEMI Patients: The SMILE Trial. J Am Coll Cardiol. 2016 Jan 26;67(3):264-72. doi: 10.1016/j.jacc.2015.10.082. PMID 26796390
- [Result] Koppara T, Joner M, Bayer G, Steigerwald K, Diener T, Wittchow E. Histopathological comparison of biodegradable polymer and permanent polymer based sirolimus eluting stents in a porcine model of coronary stent implantation. Thromb Haemost. 2012 Jun;107(6):1161-71. doi: 10.1160/TH12-01-0043. Epub 2012 Apr 26. PMID 22535188
- [Result] Koppara T, Wittchow E, Byrne RA, Bayer G, Diener T, Joner M. Permanent and biodegradable polymer coatings in the absence of antiproliferative drugs in a porcine model of coronary artery stenting. EuroIntervention. 2016 Jan 22;11(9):1020-6. doi: 10.4244/EIJY14M10_08. PMID 25317851
- [Result] Stefanini GG, Holmes DR Jr. Drug-eluting coronary-artery stents. N Engl J Med. 2013 Jan 17;368(3):254-65. doi: 10.1056/NEJMra1210816. No abstract available. PMID 23323902
- [Result] Hansson L, Hedner T, Dahlof B. Prospective randomized open blinded end-point (PROBE) study. A novel design for intervention trials. Prospective Randomized Open Blinded End-Point. Blood Press. 1992 Aug;1(2):113-9. doi: 10.3109/08037059209077502. PMID 1366259
- [Result] Stone GW, Sabik JF, Serruys PW, Simonton CA, Genereux P, Puskas J, Kandzari DE, Morice MC, Lembo N, Brown WM 3rd, Taggart DP, Banning A, Merkely B, Horkay F, Boonstra PW, van Boven AJ, Ungi I, Bogats G, Mansour S, Noiseux N, Sabate M, Pomar J, Hickey M, Gershlick A, Buszman P, Bochenek A, Schampaert E, Page P, Dressler O, Kosmidou I, Mehran R, Pocock SJ, Kappetein AP; EXCEL Trial Investigators. Everolimus-Eluting Stents or Bypass Surgery for Left Main Coronary Artery Disease. N Engl J Med. 2016 Dec 8;375(23):2223-2235. doi: 10.1056/NEJMoa1610227. Epub 2016 Oct 31. PMID 27797291
- [Derived] den Dekker WK, Elscot JJ, Bennett J, Schotborgh CE, van der Schaaf R, Sabate M, Moreno R, Ameloot K, van Bommel R, Forlani D, van Reet B, Esposito G, Dirksen MT, Ruifrok WPT, Everaert BRC, Van Mieghem C, Cummins P, Lenzen M, Brugaletta S, Boersma E, Van Mieghem NM, Diletti R; BIOVASC Investigators. Timing of Complete Multivessel Revascularization in Acute Coronary Syndrome: 2-Year Results of the BIOVASC Study. JACC Cardiovasc Interv. 2024 Dec 23;17(24):2866-2874. doi: 10.1016/j.jcin.2024.09.058. PMID 39722269
- [Derived] Diletti R, den Dekker WK, Bennett J, Schotborgh CE, van der Schaaf R, Sabate M, Moreno R, Ameloot K, van Bommel R, Forlani D, van Reet B, Esposito G, Dirksen MT, Ruifrok WPT, Everaert BRC, Van Mieghem C, Elscot JJ, Cummins P, Lenzen M, Brugaletta S, Boersma E, Van Mieghem NM; BIOVASC Investigators. Immediate versus staged complete revascularisation in patients presenting with acute coronary syndrome and multivessel coronary disease (BIOVASC): a prospective, open-label, non-inferiority, randomised trial. Lancet. 2023 Apr 8;401(10383):1172-1182. doi: 10.1016/S0140-6736(23)00351-3. Epub 2023 Mar 5. PMID 36889333
- [Derived] den Dekker WK, Van Mieghem NM, Bennett J, Sabate M, Esposito G, van Bommel RJ, Daemen J, Vrolix M, Cummins PA, Lenzen MJ, Boersma E, Zijlstra F, Diletti R; BioVasc Trial Investigators. Percutaneous complete revascularization strategies using sirolimus-eluting biodegradable polymer-coated stents in patients presenting with acute coronary syndrome and multivessel disease: Rationale and design of the BIOVASC trial. Am Heart J. 2020 Sep;227:111-117. doi: 10.1016/j.ahj.2020.06.006. Epub 2020 Jun 15. PMID 32739537
- [Derived] Kuno T, Ueyama H, Rao SV, Cohen MG, Tamis-Holland JE, Thompson C, Takagi H, Bangalore S. Percutaneous coronary intervention or coronary artery bypass graft surgery for left main coronary artery disease: A meta-analysis of randomized trials. Am Heart J. 2020 Sep;227:9-10. doi: 10.1016/j.ahj.2020.06.001. Epub 2020 Jun 7. PMID 32640370